CLINICAL TRIAL: NCT06807736
Title: PrEPared to Choose (PtC): An Implementation Study of the Delivery of Cabotegravir Long-acting Injectable Pre-exposure Prophylaxis (PrEP) as an HIV Prevention Product Option Within a PrEP Choice Context in a Real World Setting in Cape Town.
Brief Title: PrEPared to Choose (PtC) is an Implementation Study of the Delivery of Cabotegravir Long-acting, an Injectable Pre-exposure Prophylaxis (PrEP) Option for HIV Prevention. Injectable PrEP Will be Offered Alongside Oral and Vaginal Ring PrEP From Within a Real-world Context in Cape Town, South Africa.
Acronym: PtC
Status: Recruiting | Type: Observational
Sponsor: Desmond Tutu HIV Foundation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: PrEPared to Choose
Record Dates: First submitted 2025-01-14; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: HIV Infection; Sexual and Reproductive Health
Keywords: HIV prevention; Pre-exposure prophylaxis; Injectable PrEP; Adolescents and young people; South Africa; Cabotegravir long-acting; PrEP Choice
MeSH Terms: conditions — HIV Infections; Coitus | interventions — cabotegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Injectable PrEP User: Participants that select to use injectable PrEP (Cabotegravir long-acting) at baseline.
  Interventions: Drug: Cabotegravir long-acting
- Oral PrEP user: Participants that select to use oral PrEP at baseline.
  Interventions: Drug: Tenofovir emtricitabine
- Ring User: Participants that select to use vaginal ring PrEP (DapiRing) at baseline.
  Interventions: Drug: Dapivirine containing vaginal ring

INTERVENTIONS:
Drug: Cabotegravir long-acting — 3ml intramuscular injection containing 600mg of Cabotegravir
  Other Names: Apretude
  Groups: Injectable PrEP User
Drug: Tenofovir emtricitabine — Oral tablet taken daily to PrEP HIV infection.
  Groups: Oral PrEP user
Drug: Dapivirine containing vaginal ring — Intra-vaginal silicone ring containing slow-release Dapivirine, replaced every 28 days
  Groups: Ring User

SUMMARY:
The goal of this clinical trial is to offer adolescents and young people in Cape Town, South Africa different HIV pre-exposure prophylaxis (PrEP) products and describe how they use these products over an 18-month period. The study has both clinical and implementation primary aims. The primary clinical aim is short and long-term persistence on PrEP. Persistence is defined as the length of time that a participant shows continuous use of a PrEP product as intended, without stopping PrEP or switching to another PrEP product. The primary implementation aim involves the determination of factors that either enable or serve as a barrier to PrEP uptake and continuation.

Participants will be offered a choice between three antiretroviral-containing PrEP products: (1) a Tenofovir-based oral tablet that needs to be taken daily; (2) a vaginal ring containing Dapivirine that provides HIV protection for up to one month; and (3) an intramuscular injection containing Cabotegravir that provides HIV protection for up to two months. Participants will be able to use the same product throughout the study, switch between products, or stop and restart on PrEP at any point.

The study will be offered from two study sites: the first is a mobile clinic that rotates on a fixed schedule across the study area and the second is a fixed-location government primary healthcare clinic. The study will be open to confirmed HIV-negative individuals, including adolescent girls and young women (aged 15-29 years), young gender and sexually diverse populations aged 15-29 years (including men who have sex with men, transgender people, and non-binary people), and their collective sexual partners (including heterosexual, cisgender men) of any age.

DETAILED DESCRIPTION:
The PrEPared to Choose (PtC) study seeks to describe patterns of persistence on HIV pre-exposure prophylaxis (PrEP) products, individually and overall, amongst a cohort of South African adolescents and youth when offered a choice between PrEP products in real-world public health facility and mobile clinic settings. The study will further seek to understand implementation barriers and enablers in PrEP adoption (decision to use any PrEP product), initiation (first dose of any PrEP product), and persistence amongst both PrEP users (adolescents and youth) and PrEP providers (healthcare providers).

This study will utilise a prospective cohort design that recruits 1800 adolescents and young people, specifically adolescent girls and young women, including pregnant and lacting women (15-29 years), young male key populations including men who have sex with men and male sex workers (15-29 years), and their collective intimate male partners (any age).

Participants will be invited to choose to initiate on one of three types of PrEP (injectable, oral, or vaginal ring PrEP). Participants will be able to use the same product throughout the study, switch between products, or stop and restart on PrEP at any point. Participants will be followed for 7 months to meet the primary outcome of short-term persistence and for a further 18 months to meet the secondary outcome of long-term persistence. Persistence will be defined as the continuous use of the selected product as intended with (a) <7 day gap and (b) <28 day gap in PrEP availability for daily dosing (oral PrEP), vaginal ring insertion, or subsequent injection. The 7-day window aligns with previous trial definitions of on-time dosing while the 28-day window aligns with pragmatic definitions of on-time dosing for PrEP in the South African context.

The three products available will include: (1) a Tenofovir-based oral tablet that needs to be taken daily and is provided as a 30-day supply of oral tablets; (2) a intra-vaginal silicone ring containing slow-release Dapivirine that provides HIV protection for up to 28 days; and (3) an intramuscular injection containing Cabotegravir that provides HIV protection for up to two months. The study will aim to recruit up to 900 participants that initiate on injectable PrEP, up to 600 participants that initiate on oral PrEP, and up to 300 participants that initiate on vaginal ring PrEP.

PrEP choice counselling will be co-created with PrEP providers and young PrEP users (members of an existing PrEP-orientated youth reference group) and delivered by trained, adolescent-friendly HIV counsellors. PrEP will be administered by NIMART trained (Nurse Initiated Management of Anti-Retroviral Therapy) nurses at two clinical sites: a stationary government primary health care facility and a mobile clinic service that rotates on a fixed schedule through the study area. Participants will initiate at a single site but remain eligible to receive subsequent product refills/doses at the other site if desired.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be HIV negative at baseline
* All participants must have a body weight ¬> 35kg at baseline
* All participants must be older than 15 years. Specific age criteria will be applied to certain population groups.
* All participants must be currently resident in the study area
* All participants must be able to provide written, informed voluntary consent to partake in the study and willing and able to receive an injectable pre-exposure prophylaxis (PrEP) product

Exclusion Criteria:

* Confirmed HIV-positive test result and/or signs and symptoms of an acute HIV infection
* Clinical conditions contraindicated for the chosen PrEP product as per SAHPRA regulations, including use of known contraindicated medications.
* Allergy to any of the study products
* Do not spend a reasonable amount of time in the study area as residents, for school, or work, or are otherwise unable to participate in clinical or study visits for geographical reasons, according to the site investigator
* Medical, social or other condition that, in the opinion of the site investigator, would interfere with the conduct of the study or safety of the participant (e.g., provided by self-report, or found upon medical history and examination or in available medical records)
* Current enrolment in another HIV prevention clinical trial that in the opinion of the site investigator, would interfere with the conduct of the study or safety of the participant (as verified by registration on the South African Medical Research Council biometric co-enrolment prevention system).

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the Klipfontein-Mitchells Plain Health sub-district (a peri-urban, high-density, low socio-economic setting) in Cape Town, South Africa. Participants can access the study through the mobile clinic (which rotates through the study area on a fixed schedule) or a local government primary healthcare facility. The target study population includes adolescent girls and young women (aged 15 -29 years) and their intimate male partners (>15 years). Gender and sexually diverse populations, including men who have sex with men, transgender women, and transgender men, are eligible for study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Short-term persistence | 7 months
  Persistence (return for PrEP product within a scheduled visit window) over the short-term (7 months) will be measured and reported as persistent vs non-persistent continuation on each specific PrEP product (oral, injectable, ring) and on PrEP overall (accounting for continuation after switching to a different PrEP product). Non-persistence will be defined as failure to return for PrEP within (a) 7 days of the scheduled visit and (b) 28 days of the scheduled visit.
Primary implementation aim. | 7 months; 18 months
  The combination of implementation strategies best achieve pre-exposure prophylaxis (PrEP) adoption, active implementation (initiation), and persistence (sustainment) outcomes over the short term (7 months) and the long term (18 months) will be collected and reported within a RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework. This will include implementation strategies that describe PrEP choice counselling, the integration of injectable PrEP into standard of care clinical practise, and the differentiating practises required for the effective delivery of PrEP from community based and healthcare facility based settings.

SECONDARY OUTCOMES:
Durable persistence | 18 months
  Persistence (return for PrEP product within a scheduled visit window) over the long-term (18 months) will be measured and reported as persistent vs non-persistent continuation on each specific PrEP product (oral, injectable, ring) and on PrEP overall (accounting for continuation after switching to a different PrEP product). Non-persistence will be defined as failure to return for PrEP within (a) 7 days of the scheduled visit and (b) 28 days of the scheduled visit.
Time on PrEP | 18 months
  Time on PrEP based on expected (e.g. injections given; product collections as logged in dispency records) vs actual (e.g. self-reported patterns of use by the oral and ring PrEP user) PrEP coverage.
Safety of PrEP products | 18 months
  Reported frequency, timing, and nature of self reported and/or clinically identified adverse events (including clinical events, intimate partner violence, and pregnancy and infant outcomes).
Tolerability of PrEP products | 18 months
  Descriptive reports of product tolerability as per the frequency, timing, and nature of self-reported adverse side effect records. Side effects are asked about by HIV counsellors and research nurses at each study visit and rention officers during retention communications.
Acceptability of PrEP products | 18 months
  Descriptive quantitative and qualitative summaries of reasons for pre-exposure prophylaxis (PrEP) pause or discontinuation. Qualitative questionnaires and in-depth interviews that include questions on PrEP product and PrEP service acceptability are held every 6 months with a sub-set of PrEP users.
HIV testing in a context of PrEP choice | 18 months
  Sensitivity and specificity of counsellor-administered 3rd and 4th generation rapid Antigen/Antibody (Ag/Ab) HIV test compared to laboratory-based NAAT (Nucleic Acid Amplification Tests) testing results in injectable pre-exposure prophylaxis-using (Cabotegrvair long-acting initiated) participants as measured at discreet timepoints (baseline, month 1, month 7, and month 18) throughout the study.

OTHER OUTCOMES:
HIV incidence | 18 months
  HIV incidence (as determined by HIV rapid and laboratory NAAT tests at each study visit and an overview of the medical records of participants lost to follow up and its correlation with individual PrEP use patterns (including PrEP product choice, PrEP persistence, product switching, and/or PrEP pauses and discontinuation over the 18 month study period). This outcome will be reported, however, the sample size of the study is insufficient to allow for a formal analysis of HIV incidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Desmond Tutu Health Foundation, Cape Town, Western Province, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pike C, Rousseau E, Macdonald P, Mapukata P, Lebelo K, Joseph-Davey D, Little F, Bekker LG. PrEPared to choose: the protocol for an implementation study of the delivery of cabotegravir long-acting injectable pre-exposure prophylaxis (PrEP) as an HIV prevention product option within a real world PrEP choice context in cape town. BMC Public Health. 2025 Sep 24;25(1):3109. doi: 10.1186/s12889-025-24370-z. PMID 40993613